# Official Title of the study

Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Oncology Patients With Colon Cancer Undergoing Active Treatment

**NCT** 

NOT Available

# DATE OF THE DOCUMENT

01/09/2024

## TITLE:

Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Oncology Patients With Colon Cancer Undergoing Active Treatment

#### INFORMED CONSENT FORM

You are being offered the opportunity to participate in a research study titled: "Effects of a Cognitive Training Program on Chemotherapy-induced Cognitive Impairment (Chemobrain) in Oncology Patients With Colon Cancer Undergoing Active Treatment," which is being conducted by Samuel Jiménez Sánchez, a thesis student, under the direction of Eduardo José Fernández, and has been evaluated and approved by the Research Ethics Committee of SACYL.

WHAT IS THE PURPOSE OF THE STUDY? The objective of this study is to improve the quality of life of breast cancer patients through everyday cognition training, proposing an assessment and intervention based on the importance of real cognitive functioning during the resolution of complex tasks in daily life, prioritizing the improvement of autonomy, improving sleep quality and reducing anxiety.

You are being asked to participate in this study because you are an oncology patient and your cognitive functioning may be affected due to the cancer process itself or by the different treatments you are receiving.

WHAT DOES YOUR PARTICIPATION CONSIST OF? You are asked for permission to use the results regarding different indexes and scales for scientific purposes, to analyze the impact of the oncological process on the patient's cognitive performance. Participation in this project does not involve any alteration in the treatment you are undergoing.

WHAT ARE THE BENEFITS? It is very likely that the results obtained in this research will have a positive value for you, and you will also contribute to a better understanding of your situation and improve the quality of life and cognitive performance of oncology patients.

WHAT HAPPENS IF YOU DO NOT WANT TO PARTICIPATE IN THIS STUDY? Your participation in this study is entirely voluntary. If you decide not to participate in the study, this will not modify the treatment and follow-up of your situation by your doctor or the rest of the health personnel who take care of your disease. You may also answer whatever you want and you may stop the interview whenever you consider it.

**CONFIDENTIALITY** All your data, as well as all medical information related to your situation, will be treated with absolute confidentiality by the personnel in charge of the research. Likewise, if the results of the study <sup>1</sup> were to be published in scientific journals, at no time will personal data of the patients who have collaborated in this research be provided. As contemplated by Organic Law 3/2018, of December 5, on the Protection of Personal Data and Guarantee of Digital Rights, you may exercise your right to access, rectify or cancel your data by contacting the principal investigator of this study. <sup>2</sup>

### **INFORMED CONSENT**

Title of the Project: EVERYDAY COGNITION TRAINING OF BREAST CANCER PATIENTS WITHOUT COGNITIVE IMPAIRMENT

It is being carried out by Samuel Jiménez Sánchez, a thesis student, under the direction of Eduardo José Fernández, and has been evaluated and approved by the Research Ethics Committee of SACYL.

| I, | , have |
|---|---|
| been informed by | |
| collaborator of the aforementioned research project, and I declare that: | |

- I have received enough information about the study
- I have been able to ask questions about the study
- I have received satisfactory answers to my questions I understand that my participation is voluntary I understand that all my data will be treated confidentially

With this I give my consent to participate in this study,

| Date: | Date: |
|-------|--------------------------------|
| | Signature of the caregiver: |
| | Signature of the investigator: |